CLINICAL TRIAL: NCT00788307
Title: Phase I Trial of In Situ Gene Therapy for Locally Recurrent Prostate Cancer Following Radiation Therapy Failure Using Sodium/Iodide Symporter and Radioiodine
Brief Title: Gene Therapy and Radioactive Iodine in Treating Patients With Locally Recurrent Prostate Cancer That Did Not Respond to External-Beam Radiation Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: closed early due to poor accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0252; P30CA015083 (NIH); MC0252 (Other: Mayo Clinic Cancer Center); 06-009392 (Other: Mayo Clinic IRB); NCI-2009-01195 (Other: NCI-CTRP)
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triiodothyronine; Reverse Transcriptase Polymerase Chain Reaction; Iodine-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Biological: Ad5-CMV-NIS; Drug: liothyronine sodium; Genetic: reverse transcriptase-polymerase chain reaction; Other: laboratory biomarker analysis; Radiation: iodine I 131

INTERVENTIONS:
Biological: Ad5-CMV-NIS
Drug: liothyronine sodium
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis
Radiation: iodine I 131

SUMMARY:
RATIONALE: Radioactive drugs, such as radioactive iodine, may carry radiation directly to tumor cells and not harm normal cells. Placing a gene called Ad5CMV-NIS in prostate cancer cells may help the prostate cells take in more radioactive iodine and thus kill the cancer cells. Drugs, such as liothyronine sodium, may protect the thyroid from the side effects of radioactive iodine.

PURPOSE: This phase I trial is studying the side effects and best dose of gene therapy given together with radioactive iodine in treating patients with locally recurrent prostate cancer that did not respond to external-beam radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety and tolerance of Ad5CMV-NIS administered intraprostatically followed by radioiodine treatment in patients with locally recurrent adenocarcinoma of the prostate following external beam radiotherapy.
* To determine the maximum tolerated dose of Ad5CMV-NIS in these patients.

Secondary

* To evaluate the PSA response rates, duration, and time to PSA progression in these patients.
* To evaluate the immune response to Ad5CMV-NIS.

OUTLINE: This is a dose-escalation study of Ad5CMV-NIS.

Patients receive intraprostate Ad5CMV-NIS, via transperineal injection under anesthesia, on day 1. They receive dosimetry oral iodine I 123 on day 4 and undergo image studies periodically for the next 24 hours for measurement of radioiodine uptake. Patients receive therapeutic oral iodine I 131 on day 5.

All patients with intact thyroid glands (i.e., not previously surgically removed or ablated) receive TSH suppressive doses of oral liothyronine sodium 3 times daily for 10 days prior and for 15 days post administration of iodine I 123.

Blood samples are collected periodically for measurement of PSA, fT4, and TSH; and peripheral blood cells are monitored for evidence of virus DNA via quantitative reverse-transcriptase-PCR.

After completion of study therapy, patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 8 years. A transrectal tumor biopsy is to be performed at 3 months and 1 year post-treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent adenocarcinoma of the prostate within the past year

  * No transitional cell, small cell, or squamous cell carcinoma of the prostate
  * Local recurrence
* Disease recurred ≥ 18 months after completion of prior external beam radiotherapy (EBRT) for stage T1-T2b, N0/X, M0 disease

  * Biochemical failure as defined by the Phoenix definition (rise in PSA by 2 ng/mL or more above the nadir PSA)

    * PSA ≥ 0.3 ng/mL to < 20 ng/mL measured within the past 30 days
  * Pre-EBRT PSA < 50 ng/mL
  * Prior locally recurrent hormone-refractory disease allowed
* American Urologic Association Obstructive Symptom Index Score ≤ 24
* No known standard therapy that is potentially curative or definitely capable of extending life expectancy
* No evidence of or history of metastatic adenocarcinoma of the prostate

  * Negative radiographic metastatic work-up including whole-body radionuclide bone scan, CT and/or MR scan of the pelvis and abdomen, and chest x-ray

    * Patients with suspicious areas on conventional imaging studies are eligible provided they are biopsy negative
  * No known CNS metastases
* No prostate size > 140 cc

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 8.5 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* INR ≤ 1.4 times ULN
* Creatinine ≤ 1.5 times ULN
* Thyroid-stimulating hormone 0.3-5.0 uIU/mL and free thyroxine 0.8-1.87 ng/dL
* Willing to provide biologic specimens and participate in imaging studies as required
* Willing to maintain a low-iodine diet for 12 days

  * Starting 7 days prior to study virus injection continuing until after the iodine I 131 radioiodine therapy on day 5
* No more than 1 of the following renal/genitourinary toxicities:

  * Bladder spasms
  * Dysuria (painful urination)
  * Genitourinary fistula
  * Hemoglobinuria
  * Incontinence
  * Operative injury to bladder and/or ureter
  * Proteinuria
  * Renal failure
  * Uretal obstruction
  * Urinary frequency/urgency
  * Urinary retention
  * Urine color change (not related to other dietary or physiologic cause [e.g., bilirubin, concentrated urine, or hematuria])
  * Other renal/genitourinary toxicities
* No urinary tract infection within 72 hours prior to registration
* No pubic arch interference study demonstrating unacceptable prostate access by the transperineal approach
* No absence of rectum or other anatomic features that would preclude transperineal needle insertion into the prostate
* No coagulopathy that contraindicates transperineal and intraprostatic needle insertion
* No other cancer within the past 2 years, except for squamous cell and basal cell skin cancers
* No uncontrolled infection or fever > 100°F
* No known cardiac disease
* No seizure disorder
* No documented history of HIV positivity or other acquired immunodeficiency disorder or congenital immunodeficiency disorder

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from acute, reversible effects of prior chemotherapy
* Androgen-deprivation therapy (if applicable) initiated more than 3 months prior to registration

  * Patients who have undergone bilateral orchiectomy are eligible if they meet all other criteria
* At least 6 weeks since prior bicalutamide, nilutamide, or oral or intravenous iodinated contrast
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas), immunotherapy, biologic therapy, or other experimental drugs
* At least 4 weeks since prior and no concurrent anti-androgens (e.g., flutamide, estrogens, ketoconazole, PC-SPES, finasteride, or megestrol acetate)
* At least 2 weeks since prior and no concurrent exogenous corticosteroids

  * Patients clinically proven to require maintenance steroids allowed provided there has been no change in their dose within the past 6 weeks
* No antibiotic therapy within the past 72 hours
* No prior organ transplantation
* No prior salvage prostatectomy or brachytherapy
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational
* No concurrent prophylactic use of colony-stimulating factors
* No concurrent enrollment in any other study involving a pharmacologic agent (drugs, biologics, immunotherapy approaches, gene therapy) whether for symptom control or therapeutic intent

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-11-03 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Number of toxicity incidents by NCI CTCAE v3.0 criteria | 3 years

SECONDARY OUTCOMES:
Time to PSA progression | 3 years
Survival | 3 years
Incidence and duration of PSA response | 3 years
Duration of PSA control | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Davis, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials